CLINICAL TRIAL: NCT03432156
Title: Autologous Tcm Cells Immunotherapy in Patients With High-risk Recurrent Stage II Non-Small Cell Lung Cancer (NSCLC) After Postoperative Chemotherapy
Brief Title: Autologous Tcm Cells Immunotherapy in Patients With Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jing Wang, assistant director physician, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingFH-JW-180202-1
Record Dates: First submitted 2018-02-02; First posted 2018-02-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: immunotherapy; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Experimental group: immunotherapy. subjects who are treated with autologous Tcm cells immunotherapy.
  No intervention group: subjects who are treated without autologous Tcm cells immunotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): subjects who are treated with autologous Tcm cells immunotherapy
  Interventions: Biological: Autologous Tcm cells immunotherapy
- No intervention group (No Intervention): subjects who are treated without autologous Tcm cells immunotherapy

INTERVENTIONS:
Biological: Autologous Tcm cells immunotherapy — Autologous Tcm cells immunotherapy is to collect patient's own immune cells in peripheral blood and then given back to the patient after amplified in vitro.
  Arms: Experimental group

SUMMARY:
Autologous Tcm cells immunotherapy combining surgery or chemotherapy could effectively prolong survival period and improve quality of life in patients.

DETAILED DESCRIPTION:
Autologous central memory T cells (Tcm) cells immunotherapy is to collect patient's own immune cells in peripheral blood and then given back to the patient after amplified in vitro that can improve the anti-tumor immune response and is effective treatment of the cancer. Tcm cells are effective anti-tumor immune cells that exhibit the long-term survival and self-renewal capacity in vivo. Autologous Tcm cells immunotherapy combining surgery or chemotherapy could effectively prolong survival period and improve quality of life in patients.

Lung cancer is the leading cause of cancer related deaths, which account for one third of all deaths due to cancer worldwide. The most common histologic type of lung cancer is non-small-cell lung cancer (NSCLC) that is accounting for almost 85%. There are no targeted therapeutics in patients with high-risk recurrent stage II NSCLC after postoperative chemotherapy, therefore, autologous Tcm cells immunotherapy would be a safe and effective treatment.

The aim of this study is to assess the efficacy and safety of autologous Tcm cells immunotherapy in patients with high-risk recurrent stage II NSCLC after postoperative chemotherapy. Patients will be randomized 1:1 either to the experimental arm to receive 3 cycles of autologous Tcm cells immunotherapy or to the no intervention arm.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study.
2. Subjects with pathologically confirmed stage II NSCLC.
3. Subjects with stage II NSCLC had treatment with surgical resection and 4 cycles of postoperative adjuvant chemotherapy before the study.
4. Karnofsky (KPS) ≥ 60.
5. One or more Serum tumor markers such as carcinoembryonic antigen (CEA), CA125, cytokeratin-19 fragment (CYFRA21-1), neuron-specific enolase (NSE), pro-grp and angiopoietin-2 (Ang-2) are double higher than normal level or durative elevator on three consecutive tests.
6. Adequate hematologic and end-organ function.
7. Subjects who could receive treatment with at least 3 cycles of autologous Tcm cells immunotherapy.
8. Subjects must be received auxiliary examination and record these results in detail before and after immunotherapy.
9. Subjects must meet the indications for autologous Tcm cells immunotherapy.

Exclusion Criteria:

1. Subjects with lung nodules, lymph nodes, brain, liver, bone or adrenal metastasis before the study.
2. Subjects who are using immunosuppressive agents or long-term immunosuppressive agents after organ transplantation.
3. Subjects with severe abnormality of coagulation.
4. History or any evidence of hemorrhage.
5. Subjects with severe infection or high fever.
6. Subjects with severe autoimmune diseases.
7. Subjects with persistent or intractable epilepsy.
8. Subjects with merging other malignant neoplasms.
9. Subjects with mental disorder.
10. Subjects with heart, liver or kidney diseases.
11. Major surgeries except for surgical resection of NSCLC were performed in 4 weeks before the study.
12. Autologous bone marrow transplantation (ABMT) in 4 weeks before the study.
13. Concurrent treatment or treatment on another study in 4 weeks before the study.
14. Pregnancy or breast-feeding.
15. There are drug abuse, medical treatment, mental illness and social disorders that would interfere with subjects' participation, or confound the results of the trial.
16. Any condition that would interfere with or endanger the safety and compliance of subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 12 weeks
  This study will evaluate the clinical efficacy and safety of autologous Tcm cells immunotherapy in patients with high-risk recurrent stage II NSCLC after postoperative chemotherapy according to progression-free survival (PFS) .

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 weeks
  This study will evaluate the overall survival of patients after autologous Tcm cells immunotherapy according to Overall Survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No